CLINICAL TRIAL: NCT07336680
Title: Effect of Ondansetron on Patient Tolerance, Efficacy and Endoscopist Workload in Unsedated Endoscopy for Upper Gastrointestinal Bleeding
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Chief physician of Gastroenterology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ON-UGIB25
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Esophagogastroduodenoscopy; Upper Gastrointestinal Bleeding (UGIB)
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous ondansetron (Experimental)
  Interventions: Drug: intravenous ondansetron
- control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: intravenous ondansetron — Intravenous administration of 8 mg ondansetron 0.5-1h prior to endoscopic procedure and gurgle 10 ml dyclonine hydrochloride viscous solution (0.01 g/mL) 15 min prior to the endoscopic procedure.
  Arms: intravenous ondansetron
Drug: Placebo — Intravenous administration of 8 ml saline 0.5-1h prior to endoscopic procedure and gurgle 10 ml dyclonine hydrochloride viscous solution (0.01 g/mL) 15 min prior to the endoscopic procedure.
  Arms: control

SUMMARY:
The goal of this clinical trial is to evaluate whether intravenous ondansetron can improve patient tolerance and reduce discomfort during unsedated emergency esophagogastroduodenoscopy (EGD). The main questions it aims to answer are:

* Does pre-procedural administration of ondansetron improve patient cooperation during emergency EGD?
* Does it improve endoscopic field visibility and improve the success rate of initial endoscopic hemostasis？
* Does it reduce the operator's perceived workload or stress?

Researchers will compare patients who received intravenous ondansetron with patients who received placebo to see if ondansetron can reduce patient discomfort and improve patient cooperation, therefore improve the quality of the procedure.

Participants will receive either intravenous ondansetron and dyclonine hydrochloride mucilage or intravenous saline and dyclonine hydrochloride mucilage prior to the endoscopic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of suspected or confirmed upper gastrointestinal bleeding with an indication for emergent endoscopic intervention.
* Capability to provide informed consent.

Exclusion Criteria:

* Presence of any contraindication to upper gastrointestinal endoscopy.
* Concurrent severe primary diseases of the respiratory, cardio-cerebrovascular, renal, central nervous, or hematologic systems.
* Pregnancy.
* Presence of neuropsychiatric disorders, including severe depression or severe anxiety.
* Presence of a known history of cardiac arrhythmia.
* Allergic to dyclonine hydrochloride or ondansetron.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
patient cooperation | from the beginning to the end of the endoscopic procedure
  evaluated by the endoscopist in numeric rating scale, 0 stands for not good at all, 10 stands for completely satisfied.

SECONDARY OUTCOMES:
gagging intensity of patient | from the beginning to the end of the endoscopic procedure
  gagging intensity of patient evaluated by the endoscopist, in numeric rating scale, 0 means none, 10 means extremely intense.
visualization quality | During the endoscopic procedure.
  Overall endoscopic visualization was evaluated at 4 locations including (i) gastric fundus, (ii) corpus, (iii) antrum, and (iv) duodenal bulb. The score is rated in the following criteria: 0, less than 25% of the surface was visible; 1, 25%-75% visible; and 2, more than 75% visible. The total score range was 0-8.
Success rate of initial endoscopic hemostasis | from the beginning to the end of the endoscopic procedure
  the proportion of patients in each group who achieved hemostasis with a single endoscopic intervention
Proportion of patients needing repeat endoscopy within 72 hours | from the time of the endoscopic procedure to 3 days after the endoscopic procedure.
  The proportion of patients who underwent a repeat upper gastrointestinal endoscopy for suspected rebleeding within 72 hours following the completion of the initial endoscopic procedure.
Recurrence of UGIB in 7 days | from the day of the procedure to 7 days after it
  The proportion of patients in whom hemostasis was initially achieved by endoscopy, but who subsequently experienced recurrent bleeding within 7 days. Recurrent bleeding is defined by the occurrence of any of the following: hematemesis, melena, hematochezia, hemodynamic instability, or endoscopic confirmation of recurrent bleeding at the original site.
endoscopist workload | From the beginning to the end of the endoscopic procedure
  Self-assessed by the endoscopist immediately after the procedure. It is measured across six dimensions-mental demand, physical demand, temporal demand, effort, performance, and frustration/anxiety-using a 0-100 mm visual analogue scale for each, where 0 represents "very low" and 100 represents "very high".
adverse event | from the beginning of the intervention to 1 week after the endoscopic procedure.
  Any adverse medical event occurring during the endoscopic procedure, regardless of its relationship to the study medication.